CLINICAL TRIAL: NCT05032300
Title: Shear Wave Elastography Technology to Evaluate the Efficacy of ESW in the Treatment of Patients With Chronic Plantar Fasciitis,a Single-blinded Randomised Controlled Trial
Brief Title: Shear Wave Elastography Technology to Evaluate the Efficacy of ESW in the Treatment of Patients With Chronic Plantar Fasciitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Yonggang Dou, Intermediate Physiotherapist, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NFEC-202101-K9-01
Record Dates: First submitted 2021-08-24; First posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Chronic Plantar Fasciitis
Keywords: extracorporeal shock wave; chronic plantar fasciitis; elastic modulus
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Home Infusion Therapy

STUDY DESIGN:
Intervention Model Description: Test group (shock wave) chronic plantar fasciitis; Control group patients with chronic plantar fasciitis;
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- focused shockwave therapy (Active Comparator): Patients will receive 6 sessions of focused shockwave therapy.
  Interventions: Device: Focused shockwave; Other: Home therapy
- control (Active Comparator): Patients in the control group will be treated using the home therapy protocol only.
  Interventions: Other: Home therapy

INTERVENTIONS:
Device: Focused shockwave — Procedure: Focused shockwave therapy received shock wave therapy once a week: first locate, touch on the heel of the patient Tenderness points, take tenderness points as treatment points;Then ask the patient to take the lower limbs straight sitting or prone position, Target intensity will be within a range of 0.15-0.25 mJ/mm2 at maximum Hz, Total of 3000 pulses; rest for 20 minutes after the treatment
  Arms: focused shockwave therapy
Other: Home therapy — Stretching and ice massage

SUMMARY:
Inflammation of the plantar fascia is called plantar fasciitis and is common in active or overweight individuals. It can be treated conservatively or surgically. Extracorporeal shock wave therapy has shown significant efficacy in the treatment of plantar fasciitis. Repeated chronic inflammation of the plantar fascia may lead to fibrous edema, thickening and even calcification in the fascia, resulting in thickening of the plantar fascia in patients with chronic plantar fasciitis and affecting the mechanical properties of the plantar fascia (changes in elastic modulus) ). Previous studies rarely involved changes in the elasticity of the plantar fascia before and after extracorporeal shock wave treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Pain at the proximal calcaneal stop of the plantar fascia
2. The pain is severe when waking up in the morning or standing and walking after sitting for a long time, and it is slightly relieved after activities, and it will be aggravated after long walking or standing for a long time
3. Pain time> 3 months
4. Visual Scoring Scale (VAS)>4
5. The pain is tingling, sore, or burning, etc
6. There is or no tender point at the bottom of the arch of the foot
7. The patient has not undergone corticosteroid injection therapy or shock wave therapy or surgery
8. X-ray confirmed no calcaneal spurs
9. The patient agrees to participate in this study

Exclusion Criteria:

1. Suffering from calcaneal stress fracture, atrophy of fat pad, compression of the little toe abductor nerve (Baxter's nerve), tarsal tunnel syndrome, sciatica, bone or soft tissue tumor, rheumatism or rheumatoid arthritis, rigidity Those with spondylitis and infection
2. those who disagree with and do not understand the treatment methods or methods of the experiment
3. those with mental disorders

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Elastic modulus and morphology of plantar fascia lesion area | Up to six months
  Sonoelastographic changes of plantar fascia after ESWT
Reduction in pain as assessed by a 0-10 visual analogue scale (VAS) | Up to six months
  Patients can score a minimum of 0 and a maximum of 10. Getting a high score indicates a bad situation.

SECONDARY OUTCOMES:
American Society of Foot and Ankle Surgery (AOFAS) Ankle and Hindfoot Function Score | Up to six months
  The AOFAS assess pain, symptoms, activities of daily living, sports, and quality of life related to foot and ankle pain. This will be assessed on a scale of 0-100, where 100 indicates no problems and 0 indicates extreme problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital ,Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol